CLINICAL TRIAL: NCT00522093
Title: Efficacy and Safety of TJ-100 in the Treatment of Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Collaborators: Tsumura USA (Industry)
Responsible Party: Principal Investigator, Akira Horiuchi, Digestive Disease Center, Showa Inan General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-100
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TJ-100 — TJ-100 2.5g three times per day for 6 weeks

SUMMARY:
TJ-100, a Japanese herbal medicine, is clinically effective in postoperative ileus. So it may activate bowel movement. This study will test the efficacy and safety of TJ-100 in the treatment of patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* chronic constipation defined as less than 3 spontaneous bowel movement frequencies per week
* had symptoms of abdominal bloating or discomfort

Exclusion Criteria:

* mechanical bowel obstruction
* clinically systemic disease-induced constipation
* pregnancy

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Bowel movement frequency, rescue medication use, symptom assessments, bowel gas volume measurement, adverse events | baseline (4 weeks)
Bowel movement frequency, rescue medication use, symptom assessments, bowel gas volume measurement, adverse events | 6 weeks
Bowel movement frequency, rescue medication use, symptom assessments, bowel gas volume measurement, adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, M.D., Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Japan